CLINICAL TRIAL: NCT00576407
Title: Phase II Study of Thymus Transplantation in Complete DiGeorge Syndrome #668
Brief Title: Thymus Transplantation in DiGeorge Syndrome #668
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sumitomo Pharma Switzerland GmbH (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00009955; 2R01AI047040-11A2 (NIH); R56 Bridge R01AI4704011A1 (Other Grant/Funding Number: NIH American Recovery and Reinvestment Act (ARRA) of 2009); 5K12HD043494-09 (NIH); R01AI047040 (NIH); 3R56AI047040-11A1S1 (NIH); R01AI054843 (NIH); #668 (Other: Duke)
Record Dates: First submitted 2007-12-17; First posted 2007-12-19 (Estimated); Results first posted 2020-02-17 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: DiGeorge Syndrome; Complete Typical DiGeorge Anomaly
Keywords: Thymus Transplantation; DiGeorge Syndrome; Athymia; Low T cell numbers; Immunoreconstitution; Primary immunodeficiency; DiGeorge Anomaly; Complete DiGeorge; Typical DiGeorge; Cultured Thymus Tissue Implantation (CTTI)
MeSH Terms: conditions — DiGeorge Syndrome; Thymic aplasia; Primary Immunodeficiency Diseases | interventions — Drug Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cultured Thymus Tissue Implantation in Complete DiGeorge (Experimental): Participants with Complete DiGeorge Syndrome, who were eligible, received cultured thymus tissue implantation (CTTI).
  No specific dose was assigned. There was a one time administration of the cultured thymus tissue.
  Interventions: Biological: Cultured Thymus Tissue for Implantation (CTTI)

INTERVENTIONS:
Biological: Cultured Thymus Tissue for Implantation (CTTI) — Cultured thymus tissue for implantation (CTTI) (previously described as transplantation) is done using allogeneic cultured postnatal tissue from unrelated thymus donors. Thymus tissue, the thymus donor, & thymus donor's birth mother were screened for safety. Approximately 2-3 weeks post-harvest thymus slices were implanted into the recipient's quadriceps. Dose was number of grams of cultured thymus tissue divided by the recipient's weight in kilograms. Minimum dose was 4 g/m2. Maximum dose 18g/m2. At time of CTTI, a skin biopsy was obtained to look for preexisting T cells. 2-3 months post-CTTI allograft biopsy to evaluate for thymopoiesis & graft rejection. At time of biopsy, skin biopsy done to look for T cell clonal populations. Post-CTTI, subjects followed by routine research immune evaluations, using blood samples for approximately 2 years.
  Other Names: Thymus Tissue; Thymus Tissue Transplantation; Thymus Transplant; CTTI

SUMMARY:
The study purpose is to determine whether cultured thymus tissue implantation (CTTI) is effective in treating typical complete DiGeorge syndrome.

DETAILED DESCRIPTION:
There is no safe and effective treatment for DiGeorge syndrome and most patients die by the age of two. Complete DiGeorge syndrome is characterized by very low T cell or very low naïve T cell numbers. In this study, typical complete DiGeorge syndrome subjects underwent human postnatal cultured thymus tissue implantation (CTTI). Thymus tissue that would otherwise be discarded was processed and then implanted into complete DiGeorge subjects in the operating room. At the time of CTTI, a skin biopsy may have been obtained to look for any preexisting T cells. After CTTI, subjects were followed by routine research immune evaluations, using blood samples obtained approximately every 2-4 weeks. At approximately 2-3 months post-CTTI subjects underwent an open biopsy of the allograft. The biopsy was done under general anesthesia in the operating room. At the time of the graft biopsy, another skin biopsy was obtained to look for clonal populations of T cells.

The protocol aims include: assessing thymopoiesis in the allograft biopsy; assessing immunoreconstitution of complete DiGeorge syndrome subjects after postnatal allogeneic cultured thymus tissue implantation; assessing minimally invasive methods of assessing thymopoiesis (flow cytometry and polymerase chain reaction (PCR); assessing pre-implant T cells which do not proliferate in response to mitogens (focusing on NK-T cells); and, assessing cultured thymus tissue implantation safety and toxicity.

ELIGIBILITY:
Inclusion Criteria:

* The subject's parent(s) signed the ICF.
* For a diagnosis of DiGeorge Syndrome (DGS), the subject had one of the following:

  * Heart defect
  * Hypoparathyroidism
  * 22q11 hemizygosity
  * 10p13 hemizygosity
  * Coloboma, heart defect, choanal atresia, growth and development retardation, genital hypoplasia, ear anomalies/ deafness CHARGE association mutation (CHD7 deletion);
  * PHA proliferative responses less than 20-fold above background.
* Subjects with typical Complete DiGeorge Anomaly (cDGA) had to have one of the following on 2 separate occasions:
* Circulating CD3+ T cells by flow cytometry < 50/mm3 or PHA < 20-fold over background

  * If CD3+ were > 50/mm3, then CD45RA+ (cluster of differentiation 45RA) CD62L+ had to be < 50/mm3
  * Or T cell receptor rearrangement excision circles (TRECs) by PCR had to be < 100 per 100,000 CD3+ cells.
* Subjects with atypical cDGA had to have both of the following with 2 studies each:

  * Circulating CD3+ T cells by flow cytometry > 500/mm3 and CD45RA+ CD62L+ CD3+ T cells < 50/mm3 and TRECs less than 100 per 100,000 CD3+ cells.
  * T cell proliferative response to PHA more than 20-fold over background. Circulating CD3+ T cells by flow cytometry > 500/mm3 and CD45RA+ CD62L+ CD3+ T cells < 50/mm3 and TRECs less than 100 per 100,000 CD3+ cells.
  * T cell proliferative response to PHA more than 20-fold over background. While T cell response to PHA might have been seen, eligible subjects were to have no T cell proliferative response to antigens (less than 20-fold response) and were to have serious clinical problems related to immunodeficiency, such as opportunistic infection or failure to thrive.

Exclusion Criteria:

* Subjects on ventilators, with tracheostomies, with cytomegalovirus (CMV) infections, or requiring ongoing steroids could still be enrolled, but their data were to be analyzed separately
* Subjects who had heart surgery < 4 weeks prior to transplant
* Heart surgery anticipated within 3 months of the proposed time of transplantation
* Ongoing parenteral steroid therapy between enrollment and transplantation
* Present or past lymphadenopathy
* Rash associated with T cell infiltration of the dermis and epidermis
* Rejection by the surgeon or anesthesiologist as surgical candidates
* Lack of sufficient muscle tissue to accept a transplant of 4 g/m2 body surface area (BSA) of the recipient
* Prior attempts at immune reconstitution, such as bone marrow transplantation or previous thymus transplantation
* Human immunodeficiency virus (HIV) infection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 1991-10 (Actual); Primary Completion 2009-04 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Louise Markert, MD, PhD, Principal Investigator — Duke University Medical Center, Pediatrics, Allergy & Immunology
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Li B, Li J, Devlin BH, Markert ML. Thymic microenvironment reconstitution after postnatal human thymus transplantation. Clin Immunol. 2011 Sep;140(3):244-59. doi: 10.1016/j.clim.2011.04.004. Epub 2011 Apr 16. PMID 21565561
- [Background] Chinn IK, Olson JA, Skinner MA, McCarthy EA, Gupton SE, Chen DF, Bonilla FA, Roberts RL, Kanariou MG, Devlin BH, Markert ML. Mechanisms of tolerance to parental parathyroid tissue when combined with human allogeneic thymus transplantation. J Allergy Clin Immunol. 2010 Oct;126(4):814-820.e8. doi: 10.1016/j.jaci.2010.07.016. Epub 2010 Sep 15. PMID 20832849
- [Background] Chinn IK, Milner JD, Scheinberg P, Douek DC, Markert ML. Thymus transplantation restores the repertoires of forkhead box protein 3 (FoxP3)+ and FoxP3- T cells in complete DiGeorge anomaly. Clin Exp Immunol. 2013 Jul;173(1):140-9. doi: 10.1111/cei.12088. PMID 23607606
- [Result] Markert ML, Sarzotti M, Ozaki DA, Sempowski GD, Rhein ME, Hale LP, Le Deist F, Alexieff MJ, Li J, Hauser ER, Haynes BF, Rice HE, Skinner MA, Mahaffey SM, Jaggers J, Stein LD, Mill MR. Thymus transplantation in complete DiGeorge syndrome: immunologic and safety evaluations in 12 patients. Blood. 2003 Aug 1;102(3):1121-30. doi: 10.1182/blood-2002-08-2545. Epub 2003 Apr 17. PMID 12702512
- [Result] Markert ML, Devlin BH, Alexieff MJ, Li J, McCarthy EA, Gupton SE, Chinn IK, Hale LP, Kepler TB, He M, Sarzotti M, Skinner MA, Rice HE, Hoehner JC. Review of 54 patients with complete DiGeorge anomaly enrolled in protocols for thymus transplantation: outcome of 44 consecutive transplants. Blood. 2007 May 15;109(10):4539-47. doi: 10.1182/blood-2006-10-048652. Epub 2007 Feb 6. PMID 17284531
- [Result] Markert ML, Devlin BH, McCarthy EA. Thymus transplantation. Clin Immunol. 2010 May;135(2):236-46. doi: 10.1016/j.clim.2010.02.007. Epub 2010 Mar 16. PMID 20236866
- [Result] Markert ML and Devlin BH. Thymic reconstitution (in Rich RR, Shearer WT, Fleischer T, Schroeder HW, Weyand CM, Frew A, eds., Clinical Immunology 3rd edn., Elsevier, Edinburgh) p 1253-1262, 2008.
- [Result] Chinn IK, Devlin BH, Li YJ, Markert ML. Long-term tolerance to allogeneic thymus transplants in complete DiGeorge anomaly. Clin Immunol. 2008 Mar;126(3):277-81. doi: 10.1016/j.clim.2007.11.009. Epub 2007 Dec 26. PMID 18155964
- [Result] Markert ML, Li J, Devlin BH, Hoehner JC, Rice HE, Skinner MA, Li YJ, Hale LP. Use of allograft biopsies to assess thymopoiesis after thymus transplantation. J Immunol. 2008 May 1;180(9):6354-64. doi: 10.4049/jimmunol.180.9.6354. PMID 18424759
- [Result] Hudson LL, Louise Markert M, Devlin BH, Haynes BF, Sempowski GD. Human T cell reconstitution in DiGeorge syndrome and HIV-1 infection. Semin Immunol. 2007 Oct;19(5):297-309. doi: 10.1016/j.smim.2007.10.002. Epub 2007 Nov 26. PMID 18035553
- [Result] Markert ML, Devlin BH, Chinn IK, McCarthy EA, Li YJ. Factors affecting success of thymus transplantation for complete DiGeorge anomaly. Am J Transplant. 2008 Aug;8(8):1729-36. doi: 10.1111/j.1600-6143.2008.02301.x. Epub 2008 Jun 28. PMID 18557726
- [Result] Markert ML, Devlin BH, Chinn IK, McCarthy EA. Thymus transplantation in complete DiGeorge anomaly. Immunol Res. 2009;44(1-3):61-70. doi: 10.1007/s12026-008-8082-5. PMID 19066739
- [Result] Markert ML, Marques JG, Neven B, Devlin BH, McCarthy EA, Chinn IK, Albuquerque AS, Silva SL, Pignata C, de Saint Basile G, Victorino RM, Picard C, Debre M, Mahlaoui N, Fischer A, Sousa AE. First use of thymus transplantation therapy for FOXN1 deficiency (nude/SCID): a report of 2 cases. Blood. 2011 Jan 13;117(2):688-96. doi: 10.1182/blood-2010-06-292490. Epub 2010 Oct 26. PMID 20978268
- [Result] Markert ML, Devlin BH, McCarthy EA, Chinn IK, Hale LP. Thymus Transplantation in Thymus Gland Pathology: Clinical, Diagnostic, and Therapeutic Features. Eds Lavinin C, Moran CA, Morandi U, Schoenhuber R. Springer-Verlag Italia, Milan, 2008, pp 255-267.

RESULTS

PARTICIPANT FLOW:
Groups:
- Cultured Thymus Tissue Implantation: Cultured Thymus Tissue Implantation (previously described as transplantation) is done using allogeneic cultured postnatal tissue from unrelated donors.
Period: Overall Study
Arm/Group | Cultured Thymus Tissue Implantation
Started | 26
Completed | 18
Not Completed | 8
Not completed — Death | 7
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Of the 26 participants enrolled, two subjects did not have cDGA (1 severe combined immunodeficiency [SCID] and 1 FoxN1) underwent cultured thymus tissue implantation as enrollment exceptions. The FoxN1 participant is included in the efficacy analysis set, thus n=25. The SCID participant is not included in the efficacy analysis set.
Groups:
- Cultured Thymus Tissue Implantation: Cultured Thymus Tissue Implantation is done using allogeneic cultured postnatal thymus tissue from unrelated donors.
Arm/Group | Cultured Thymus Tissue Implantation
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 26
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: days] | 153 (102)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Survival at 1 Year Post-Cultured Thymus Tissue Implantation (CTTI)
Description: Survival at 1 year post CTTI was assessed using the Kaplan Meier Estimated Survival. This mathematical function estimates the survival for a certain length of time.
Time Frame: 1 year post-CTTI
Population: Of the 26 participants, 2 subjects did not have cDGA (1 SCID and 1 FoxN1) and underwent CTTI as enrollment exceptions. The FoxN1 participant is included in the efficacy analysis, thus n=25. The SCID participant is not included in the efficacy analysis as CTTI cannot lead to T cell development in SCID.
Measure: Number (95% Confidence Interval); unit: % of participants who survive to 1 year
Arm/Group | Cultured Thymus Tissue Implantation
Number analyzed (Participants) | 25
% of participants who survive to 1 year | 72 [50.1 to 85.5]

2. Secondary Outcome: Survival at 2 Years Post-CTTI
Description: Survival at 2 years post CTTI was assessed using the Kaplan Meier Estimated Survival. This mathematical function estimates the survival for a certain length of time.
Time Frame: 2 years post-CTTI
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % of participants who survive to 2 years
Arm/Group | Cultured Thymus Tissue Implantation
Number analyzed (Participants) | 25
% of participants who survive to 2 years | 72 [50.1 to 85.5]

3. Secondary Outcome: Immune Reconstitution Efficacy - Total CD3 T Cells
Description: The development of total CD3 T cells at one year as measured using flow cytometry
Time Frame: 1 year post-CTTI
Population: Data were only included on cDGA and FoxN1 participants for the 1 year time point if a CD3 T cell count was performed in the relevant time period.
Measure: Median (Full Range); unit: cells/mm3
Arm/Group | Cultured Thymus Tissue Implantation
Number analyzed (Participants) | 17
cells/mm3 | 770 [182 to 1698]

4. Secondary Outcome: Immune Reconstitution Efficacy - Total CD4 T Cells
Description: The development of total CD4 T cells at one year as measured using flow cytometry
Time Frame: 1 year post-CTTI
Population: Data were only included on cDGA and FoxN1 participants for the 1 year time point if a CD4 T cell count was performed in the relevant time period.
Measure: Median (Full Range); unit: cells/mm3
Groups:
- Cultured Thymus Tissue Implantation: Cultured Thymus Tissue Implantation (previously described as transplantation)is done using allogeneic cultured postnatal tissue from unrelated donors.
Arm/Group | Cultured Thymus Tissue Implantation
Number analyzed (Participants) | 17
cells/mm3 | 570 [156 to 1376]

5. Secondary Outcome: Immune Reconstitution Efficacy - Total CD8 T Cells
Description: The development of total CD8 T cells at one year as measured using flow cytometry
Time Frame: 1 year post-CTTI
Population: Data were only included on cDGA and FoxN1 participants for the 1 year time point if a CD8 T cell count was performed in the relevant time period.
Measure: Median (Full Range); unit: cells/mm3
Arm/Group | Cultured Thymus Tissue Implantation
Number analyzed (Participants) | 16
cells/mm3 | 122 [14 to 382]

6. Secondary Outcome: Immune Reconstitution Efficacy - Naive CD4 T Cells
Description: The development of naive CD4 T cells at one year as measured using flow cytometry
Time Frame: 1 year post-CTTI
Population: Data were only included on cDGA and FoxN1 participants for the 1 year time point if a T cell count was performed in the relevant time period.
Measure: Median (Full Range); unit: cells/mm3
Arm/Group | Cultured Thymus Tissue Implantation
Number analyzed (Participants) | 13
cells/mm3 | 270 [48 to 669]

7. Secondary Outcome: Immune Reconstitution Efficacy - Naive CD8 T Cells
Description: The development of naive CD8 T cells at one year as measured using flow cytometry
Time Frame: 1 year post-CTTI
Population: as for outcome 6
Measure: Median (Full Range); unit: cells/mm3
Arm/Group | Cultured Thymus Tissue Implantation
Number analyzed (Participants) | 11
cells/mm3 | 65 [2.7 to 188]

8. Secondary Outcome: Immune Reconstitution Efficacy - Response to Mitogens
Description: The development of a T cell proliferative response to the mitogen phytohemagglutinin.
Time Frame: 1 year post-CTTI
Population: Data were only included on cDGA and FoxN1 participants for the 1 year time point if testing was performed in the relevant time period.
Measure: Median (Full Range); unit: counts/minute (cpm)
Arm/Group | Cultured Thymus Tissue Implantation
Number analyzed (Participants) | 13
counts/minute (cpm) | 133000 [53913 to 390546]

9. Secondary Outcome: Thymus Allograft Biopsy
Description: Evidence, on biopsy of the thymus tissue implanted in muscle, that shows the development of new T cells.
Time Frame: 2 to 3 months post-CTTI
Population: Data were only included on cDGA and FoxN1 participants if the participant had a biopsy of the thymus tissue implanted.
Measure: Count of Participants; unit: Participants
Arm/Group | Cultured Thymus Tissue Implantation
Number analyzed (Participants) | 19
Participants
  Evidence of thymopoiesis | 17
  Evidence of rejection | 1
  Inconclusive for thymopoiesis | 1

ADVERSE EVENTS:
Time Frame: 2 years post-CTTI
Description: Adverse events reporting on all participants (cDGA, FoxN1, and SCID) who underwent cultured thymus tissue implantation (previously described as transplantation).
Arm/Group | Cultured Thymus Tissue Implantation
All-Cause Mortality (participants affected / at risk) | 7/26
Serious Adverse Events (participants affected / at risk) | 23/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cultured Thymus Tissue Implantation (N=26)
Device related infection (Infections and infestations) | 10 (19)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pyrexia (General disorders) | 3 (3)
Staphylococcal bacteraemia (Infections and infestations) | 3 (3)
Hypotension (Vascular disorders) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (4)
Diarrhoea (Gastrointestinal disorders) | 2 (3)
Sepsis (Infections and infestations) | 2 (3)
Hypothyroidism (Endocrine disorders) | 2 (2)
Hypersensitivity (Immune system disorders) | 2 (2)
Enterococcal sepsis (Infections and infestations) | 2 (2)
Gastroenteritis rotavirus (Infections and infestations) | 2 (2)
Influenza (Infections and infestations) | 2 (2)
Parainfluenzae virus infection (Infections and infestations) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2)
Seizure (Nervous system disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonia klebsiella (Infections and infestations) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Cyanosis (Cardiac disorders) | 1 (1)
Right ventricular hypertension (Cardiac disorders) | 1 (1)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Graft versus host disease in skin (Immune system disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Croup infectious (Infections and infestations) | 1 (1)
Cystitis escherichia (Infections and infestations) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 1 (1)
Gastroenteritis adenovirus (Infections and infestations) | 1 (1)
Gastroenteritis enteroviral (Infections and infestations) | 1 (1)
Klebsiella sepsis (Infections and infestations) | 1 (1)
Lower respiratory tract infection bacterial (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 1 (1)
Pseudomonal bacteraemia (Infections and infestations) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 1 (1)
Urinary tract infection viral (Infections and infestations) | 1 (1)
Varicella (Infections and infestations) | 1 (1)
Viraemia (Infections and infestations) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Feeding intolerance (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1)
Central nervous system haemorrhage (Nervous system disorders) | 1 (1)
Cranial nerve disorder (Nervous system disorders) | 1 (1)
Febrile convulsion (Nervous system disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1)
Hypertonia (Nervous system disorders) | 1 (1)
Hypocalcaemic seizure (Nervous system disorders) | 1 (1)
Infantile spasms (Nervous system disorders) | 1 (1)
Motor dysfunction (Nervous system disorders) | 1 (1)
Glomerulonephritis minimal lesion (Renal and urinary disorders) | 1 (1)
Alveolar lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cultured Thymus Tissue Implantation (N=26)
Pyrexia (General disorders) | 15 (26)
Rash (Skin and subcutaneous tissue disorders) | 9 (17)
Device related infection (Infections and infestations) | 5 (11)
Oropharyngeal candidiasis (Infections and infestations) | 5 (6)
Alanine aminotransferase increased (Investigations) | 5 (6)
Hydronephrosis (Renal and urinary disorders) | 5 (6)
Hepatomegaly (Hepatobiliary disorders) | 5 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Staphylococcal bacteraemia (Infections and infestations) | 4 (8)
Aspartate aminotransferase increased (Investigations) | 4 (5)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4)
Hypothyroidism (Endocrine disorders) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 4 (4)
Clostridium difficile colitis (Infections and infestations) | 4 (4)
Eye infection staphylococcal (Infections and infestations) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 3 (4)
Urinary tract infection enterococcal (Infections and infestations) | 3 (4)
Eosinophilia (Blood and lymphatic system disorders) | 3 (3)
Lymphadenopathy (Blood and lymphatic system disorders) | 3 (3)
Umbilical hernia (Gastrointestinal disorders) | 3 (3)
Hypersensitivity (Immune system disorders) | 3 (3)
Ear infection (Infections and infestations) | 3 (3)
Eye infection bacterial (Infections and infestations) | 3 (3)
Gastrointestinal viral infection (Infections and infestations) | 3 (3)
Otitis media (Infections and infestations) | 3 (3)
Urinary tract infection fungal (Infections and infestations) | 3 (3)
Hypertension (Vascular disorders) | 3 (3)
Cystitis klebsiella (Infections and infestations) | 2 (4)
Candiduria (Infections and infestations) | 2 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 (2)
Splenomegaly (Blood and lymphatic system disorders) | 2 (2)
Bundle branch block right (Cardiac disorders) | 2 (2)
Hydrocele (Congenital, familial and genetic disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Pancreatic insufficiency (Gastrointestinal disorders) | 2 (2)
Generalised oedema (General disorders) | 2 (2)
Enterococcal bacteraemia (Infections and infestations) | 2 (2)
Lower respiratory tract infection bacterial (Infections and infestations) | 2 (2)
Pneumonia staphylococcal (Infections and infestations) | 2 (2)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2)
Occult blood positive (Investigations) | 2 (2)
Prothrombin time prolonged (Investigations) | 2 (2)
Feeding intolerance (Metabolism and nutrition disorders) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2)
Nephrocalcinosis (Renal and urinary disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rales (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes